CLINICAL TRIAL: NCT01110928
Title: A Multicentre, Open Label, Observational, Non-interventional Study to Evaluate on Long-term Safety and Efficacy of Norditropin® Formulation in Patients With SGA Short Stature Without Closure of Epiphyseal Discs
Brief Title: Observational Study of the Safety and Efficacy of Norditropin® in Patients With SGA (Small for Gestational Age) Short Stature That Are Still Growing
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-3812; U1111-1114-6280 (Other: WHO); JapicCTI-101123 (Registry Identifier: JAPIC)
Record Dates: First submitted 2010-04-19; First posted 2010-04-27 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Norditropin®
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Norditropin® (somatropin) prescribed at the discretion of the physician according to normal clinical practice. Safety and effectiveness data is recorded by the physician, at study initiation and every 6 months until last visit.

SUMMARY:
This study is conducted in Japan. The aim of this observational study is to collect information about the safety and efficacy of Norditropin® in the long-term treatment of patients with a SGA (small for gestational age) short stature where the growth plate in the long bones (epiphyseal disc) is not closed. An extension to the GHLIQUID-1517 trial (NCT00184717).

ELIGIBILITY:
Inclusion Criteria:

* Participation in the GHLIQUID-1517 trial
* Patients with SGA (small for gestational age) short stature that are still growing

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products
* Diabetes Mellitus
* Patients with malignant tumor(s)
* Pregnant or likely to get pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with SGA short stature that are still growing, who will either receive Norditropin® (somatropin) treatment or completed the GHLIQUID-1517 trial.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2009-11-26 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Number and type of suspected serious adverse drug reactions (SADRs) during the study period | evaluated binannually for 9 years

SECONDARY OUTCOMES:
Number of glucose intolerance events during the study period | evaluated biannually for 9 years
Adult height | Fulfilment will be evaluated once a year. Height when closure of ephiphyseal discs exists or when accomplished adult height is confirmed by physician

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Background] Toshiaki Tanaka et al, The effect of growth hormone treatment on age and height at puberty onset in short Japanese children born small for gestational age: interim analysis of Norditropin post-marketing study; Japan, Journal of Japanese Association for Human Auxology; 2017: Vol 23 No. 2 : p59
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com